CLINICAL TRIAL: NCT07390669
Title: OptimAIR: Towards Right Care in Asthma Through Point-of-care Phenotyping, Guideline-based Assessment and Management Optimalisation Using the AsthmaOptimiser in Primary Care
Acronym: OptimAIR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Practitioners Research Institute (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GPRi-2024-004; EUPAS1000000559 (Other: EU PAS Register)
Record Dates: First submitted 2026-01-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Asthma Control
Keywords: Asthma control; Primary care; ORACLE; FeNO; Oscillometry; ACQ; Blood Eosinophils; Spirometry
MeSH Terms: conditions — Cardiomyopathy, Dilated, 1C

STUDY DESIGN:
Intervention Model Description: Participants undergo one structured asthma assessment in primary care using the AsthmaOptimiser with point-of-care phenotyping (e.g., ACQ-6/CAAT, oscillometry/spirometry, FeNO, point-of-care blood eosinophils as applicable). A report with guideline-based management opportunities is provided. Participants then complete remote follow-up questionnaires via the respiratory registry at 3 and 6 months (and ACQ-6/CAAT at ~12 weeks per protocol endpoints).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OptimAIR structured asthma assessment (Experimental): Participants undergo a single structured asthma assessment in primary care using the AsthmaOptimiser with point-of-care phenotyping, followed by remote follow-up questionnaires.
  Interventions: Behavioral: AsthmaOptimiser-supported structured asthma review

INTERVENTIONS:
Behavioral: AsthmaOptimiser-supported structured asthma review — Participants receive a structured, guideline-based asthma assessment during a single study visit in primary care using the AsthmaOptimiser decision-support tool. The assessment includes patient-reported outcomes (ACQ-6, CAAT), lung function testing (oscillometry and/or spirometry), and point-of-care phenotyping (e.g., FeNO and blood eosinophils, where applicable). Based on these assessments, a report is generated summarizing asthma control, exacerbation risk, and guideline-based opportunities for treatment and management optimization. Treatment decisions remain at the discretion of the treating healthcare professional. Participants complete follow-up questionnaires via a respiratory registry at approximately 3 and 6 months after the visit.

SUMMARY:
Asthma is mainly managed in primary care, yet disease control remains suboptimal. Many patients experience ongoing symptoms, exacerbations, and frequent short-acting β₂-agonist use, while underestimating the severity of their condition. Approximately 40% of patients have uncontrolled asthma based on Asthma Control Questionnaire scores. This highlights the need for structured assessment of asthma control, risk factors, inhaler technique, and alignment of treatment with international guidelines.

Structured asthma reviews and digital support tools may help optimize and personalize asthma management, particularly for patients at increased risk of exacerbations. Novel risk prediction tools using biomarkers such as FeNO and blood eosinophils show promise but are not yet routinely used in primary care.

This study aims to assess asthma control, identify patients at higher risk of exacerbations, and explore opportunities for management optimization in primary care. In addition, it supports the development of a longitudinal respiratory registry to facilitate clinical research and participation in future clinical trials.

DETAILED DESCRIPTION:
Patients with respiratory diseases, including asthma, are predominantly managed in primary care, particularly those who have not yet experienced frequent exacerbations. Despite this, asthma control remains suboptimal in a substantial proportion of patients. Ongoing symptoms, exacerbations, and overuse of short-acting β₂-agonists (SABA) are common, and approximately 40% of patients have an Asthma Control Questionnaire (ACQ) score greater than 1.5, indicating uncontrolled asthma. In addition, patients often underestimate the severity of their disease and perceive their asthma as controlled despite persistent symptoms and exacerbations. This creates a gap between perceived and actual disease control and highlights the need for structured assessment and management.

Improved asthma care requires systematic evaluation of asthma control, future risk, trigger avoidance, inhaler technique, and appropriate pharmacological treatment in accordance with current international guidelines, such as those from the Global Initiative for Asthma (GINA). Structured asthma reviews may help identify opportunities for more personalized management and treatment optimization. Digital decision-support tools, such as the previously developed AsthmaOptimiser, can support healthcare professionals during asthma consultations and facilitate guideline-based treatment decisions.

Special attention is warranted for patients at increased risk of poor asthma outcomes, particularly exacerbations. Novel risk prediction tools, including the Oxford asthma attack risk scale (ORACLE), may help identify such patients. The ORACLE score incorporates biomarkers such as fractional exhaled nitric oxide (FeNO) and blood eosinophil counts. However, these biomarkers are not yet routinely assessed in primary care, and further research is needed to evaluate their feasibility, applicability, and added value in this setting.

In parallel, multiple new pharmacological treatment classes for respiratory diseases are under development after decades of limited innovation. The evaluation of these therapies requires large clinical trials with substantial patient participation. As most patients with respiratory diseases are treated in primary care, this setting represents a large potential pool of trial participants who may benefit from participation but are often unaware of available research opportunities.

In this context, the proposed study aims to provide insight into the prevalence of controlled and uncontrolled asthma in primary care, identify opportunities for management optimization, and explore disease phenotypes and treatable traits, particularly in patients at high risk of exacerbations. In addition, the study supports the establishment of the GPRI Respiratory Registry, which will collect up-to-date longitudinal data from patients with respiratory diseases. This registry is intended to facilitate recruitment for future research studies, address relevant scientific questions, and potentially lower barriers for patient participation in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Documented physician diagnosis of asthma
* Treated with ICS+LABA
* 1 or more exacerbation(s) requiring oral or systemic corticosteroids for at least 3 days or hospital admission, or emergency room visit within 12 months prior to the OptimAIR study visit

Exclusion Criteria:

* Well controlled asthma, defined as ACQ-6 score ≤ 0.75 and normal oscillometry (ALDS result: "normal lung function")
* Not able to understand the patient information sheet and informed consent form
* Other significant respiratory disease than asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number and distribution of identified opportunities for treatment and management optimisation (GINA-guided) | During the study visit (baseline; single visit)
  Number and distribution of guideline-based opportunities to optimise asthma treatment and management identified by the AsthmaOptimiser, based on Global Initiative for Asthma (GINA) guidance.

SECONDARY OUTCOMES:
Management changes following assessment with AsthmaOptimiser and ORACLE | From baseline to 12 weeks (follow-up via Respiratory Registry)
  Number and type of management changes following the structured assessment, including:
  1. Number and type of changes made to inhaled medication
  2. Number of inhaler device changes based on inhaler technique optimisation
  3. Number and type of lifestyle recommendations (e.g. smoking cessation)
Medium-term asthma control after assessment with AsthmaOptimiser | Baseline and 12 weeks
  Change from baseline in asthma control and health status assessed by Chronic Airways Assessment Test (CAAT) score, minimum = 0, maximum = 40, higher score means worse health status.
Medium-term asthma control after assessment with AsthmaOptimiser | Baseline and 12 weeks
  Change from baseline in asthma control and health status assessed by Asthma Control Questionnaire-6 (ACQ-6) score, minimum = 0, maximum = 6, higher score means poorer asthma control.

OTHER OUTCOMES:
Population risk for future exacerbations according to ORACLE | During the study visit (baseline; full visit participants)
  Distribution of Oxford Asthma Attack Risk Scale (ORACLE) risk scores among participants in whom the ORACLE score is calculated, it is a risk prediction model estimating the likelihood of future asthma attacks based on multiple clinical variables and biomarkers. A higher risk estimate is a worse outcome, so a greater likelihood of future asthma attacks.
Willingness to participate in future interventional clinical trials following an OptimAIR visit | Baseline + 3-months follow-up questionnaire
  Engagement with clinical trials assessed as participants' willingness to participate in an interventional clinical trial if approached during or following the OptimAIR visit
Impact of OptimAIR participation on engagement with clinical trials | 12 weeks
  Outcomes related to engagement with clinical trials (Willingness to participate in interventional clinical trials when approached through the OptimAIR visit)
Change in CAAT score in trial-eligible participants who participate in a clinical trial compared with non-participants | Baseline to 6 months follow-up
  Engagement with clinical trials assessed as change in CAAT score from baseline to 6 months in participants who are eligible for an interventional clinical trial and who choose to participate, compared with eligible participants who do not participate.

CONTACTS AND LOCATIONS:
Locations (3):
- Multiple primary care sites, Buenos Aires, Argentina
- Multiple primary care sites, Santiago, Chile
- Multiple primary care sites, Palma de Mallorca, Spain

IPD SHARING:
Plan to Share IPD: No